CLINICAL TRIAL: NCT01600352
Title: To Evaluate the Clinical Utility of Specific Autoantibody Testing in Patients With Interstitial Lung Disease
Brief Title: Specific Autoantibody Testing in Patients With Interstitial Lung Disease
Status: Completed | Type: Observational
Sponsor: Singapore General Hospital (Other)
Responsible Party: Sponsor
Other Study IDs: 2012/245/Cautoantibodies
Record Dates: First submitted 2012-05-15; First posted 2012-05-17 (Estimated); Last update posted 2017-11-08 (Actual); Status verified 2017-11

CONDITIONS: Interstitial Lung Disease
Keywords: interstitial lung disease; idiopathic pulmonary fibrosis
MeSH Terms: conditions — Lung Diseases, Interstitial; Idiopathic Pulmonary Fibrosis

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — Blood
Oversight: Data Monitoring Committee: No

SUMMARY:
The purpose of this study is to evaluate the clinical utility of specific autoantibody testing in unmasking an underlying connective tissue disorder in patients who present with interstitial lung disease and found to have weak positive ANA (1:400 titre) with no overt connective tissue disease manifestations OR borderline/negative ANA with some clinical suggestion of connective tissue disease.

DETAILED DESCRIPTION:
It has been well established that patients with connective tissue disease associated interstitial lung disease respond better to immunosuppressive therapy, and have a better outcome compared to patients with idiopathic interstitial pneumonias. This makes it imperative to identify this group of patients for management and prognostication. Unfortunately some of these patients do not demonstrate overt clinical manifestations of connective tissue disease and our current available autoantibody screen does not detect all potential autoantibodies present. We would like to test for specific autoantibodies in this group of patients to evaluate its clinical utility in identifying covert connective tissue diseases associated with interstitial lung disease.

ELIGIBILITY:
Inclusion Criteria:

1. Patients 21 years old and older
2. Patients with interstitial lung disease who have been found to have weak positive ANA (1:400 titre) with no overt connective tissue disease manifestations OR borderline/negative ANA with some clinical suggestion of connective tissue disease will be offered specific autoantibody testing

Exclusion Criteria:

1. Inability and unwillingness to sign informed consent
2. Patients who are pregnant or have underlying malignancy

Ages: 21 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with weak positive ANA (1:400 titre) and no overt connective tissue disease manifestations OR borderline/negative ANA with some clinical suggestion of connective tissue disease.
Sampling Method: Non-Probability Sample
Enrollment: 20 (Actual)
Dates: Start 2012-05; Primary Completion 2017-04 (Actual); Study Completion 2017-04 (Actual)

PRIMARY OUTCOMES:
Clinical utility of specific autoantibody testing | 3 months
  Utility of specific autoantibodies to diagnose underlying connective tissue disease in patients presenting with interstitial lung disease who do not demonstrate overt clinical manifestations of connective tissue disease and our current available autoantibody screen does not detect all potential autoantibodies present.

CONTACTS AND LOCATIONS:
Overall Officials: Su Ying Low, BMBCh, Principal Investigator — Singapore General Hospital
Locations (1):
- Singapore General Hospital, Singapore, Singapore

REFERENCES:
- [Background] de Lauretis A, Veeraraghavan S, Renzoni E. Review series: Aspects of interstitial lung disease: connective tissue disease-associated interstitial lung disease: how does it differ from IPF? How should the clinical approach differ? Chron Respir Dis. 2011;8(1):53-82. doi: 10.1177/1479972310393758. PMID 21339375
- [Background] Friedman AW, Targoff IN, Arnett FC. Interstitial lung disease with autoantibodies against aminoacyl-tRNA synthetases in the absence of clinically apparent myositis. Semin Arthritis Rheum. 1996 Aug;26(1):459-67. doi: 10.1016/s0049-0172(96)80026-6. PMID 8870113
- [Background] Corte TJ, Copley SJ, Desai SR, Zappala CJ, Hansell DM, Nicholson AG, Colby TV, Renzoni E, Maher TM, Wells AU. Significance of connective tissue disease features in idiopathic interstitial pneumonia. Eur Respir J. 2012 Mar;39(3):661-8. doi: 10.1183/09031936.00174910. Epub 2011 Sep 15. PMID 21920896
- [Background] Fischer A, West SG, Swigris JJ, Brown KK, du Bois RM. Connective tissue disease-associated interstitial lung disease: a call for clarification. Chest. 2010 Aug;138(2):251-6. doi: 10.1378/chest.10-0194. PMID 20682528